CLINICAL TRIAL: NCT02550002
Title: Comparison of Treatment rOutine Using afLibERcept: Strict vs relAxed retreatmeNT Regimen (TOLERANT Study)
Brief Title: Comparison of Treatment rOutine Using afLibERcept: Strict vs relAxed retreatmeNT Regimen
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: TOLERANT
Record Dates: First submitted 2015-09-01; First posted 2015-09-15 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Strict treatment regimen with aflibercept: Treatment intervals with aflibercept in the strict retinal fluid treatment regimen will be extended by two weeks only if no SRF in the central subfoveal field and no IRF can be detected SD-OCT examination.
  Interventions: Drug: Aflibercept
- Relaxed treatment regimen with aflibercept: Treatment intervals with aflibercept in the relaxed retinal fluid treatment regimen will be extended by two weeks only if SRF in the central subfoveal field is ≤100 μm in a vertical extent and no IRF is detected on SD-OCT examination.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea

SUMMARY:
The primary objective of this study is to test non-inferiority of aflibercept "treat and extend" using a relaxed retinal fluid management relative to aflibercept "treat and extend" using a strict retinal fluid management SD-OCT (spectral domain optical coherence tomography) disease activity guided retreatment with respect to best-corrected visual acuity (BCVA) from baseline to end of treatment.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of blindness in the elderly population in developed countries. Severe visual loss in AMD usually occurs in patients with neovascular AMD (nAMD), which is caused by vascular endothelial growth factor A (VEGF-A) driven choroidal neovascularization (CNV).

Intravitreal therapy with VEGF-A inhibitors is the current standard treatment for nAMD. Optimization of current VEGF-A therapies includes finding a dosing regimen that maximizes visual acuity (VA) and minimizes the frequency of intravitreal injections and associated risks of treatment.

The "treat and extend" protocol is OCT guided with the primary aim of complete resolution of all retinal fluid, i.e. both intraretinal fluid (IRF) and subretinal fluid (SRF), both of which are considered to be a sign of disease activity. Once all fluid is resolved, an extension of the treatment interval by 2 weeks is mandated. If there is return of either SRF or IRF, the interval is shortened by one week. Currently, the relevance of both IRF and SRF in relation to best-corrected visual acuity (BCVA) outcomes is still being disputed. From the CATT and VIEW studies there is some reason to suspect that some SRF may be allowed to remain to extend the treatment interval without affecting BCVA. In contrast to IRF which has clearly been shown to correlate with poorer VA and is considered to be a sign of active disease, SRF may only be a sign of impaired pumping function of the RPE, similar to what is seen in central serous chorioretinopathy and as such may not be considered as an indication of ongoing disease activity. The consequence of insisting upon complete lack of SRF (strict approach) is more injections and therefore increased exposure of the retina to anti-VEGF agents. And there are recent reports that frequent intravitreal injections may lead to changes in the retinal nerve fiber layer and increased risk of geographic atrophy development. As a consequence, limiting the number of injections would be desirable if the same VA result could be achieved. From the pivotal anti-VEGF studies it has become apparent that patients show an individualised response to therapy. As such optimization of individualized treatment needs to be explored and understood. This study aims to explore further the "treat and extend" approach and will evaluate and compare two individualized aflibercept treatment regimens, differentiated by the definition of disease activity which determines the treatment interval until the next injection. The aim will be to determine whether small amounts of SRF may be tolerated using a "treat and extend" regimen in the treatment of nAMD and whether the presence and extent of both intra-retinal fluid and/or sub-retinal fluid (SRF) helps to decide on extension or reduction of treatment intervals in a "treat and extend" regimen. The results will be used to generate further recommendations about strict versus relaxed treatment approaches and how they can be utilised within a clinically practical "treat and extend" approach to maximize patient outcomes, while reducing the need for potentially unnecessary intravitreal injections.

Taking all together, the study aims for optimization of flexible patient treatment.

ELIGIBILITY:
Inclusion Criteria:

General:

* Informed consent as documented by signature of the patient on the informed consent form.
* Male or female, ≥50 years of age.

Study eye:

* Diagnosis ofl CNV secondary to wAMD without restriction of lesion size, with visual impairment due to an active wAMD lesion. Active wAMD lesions are characterised by the following:

  * Evidence of SRF and/or IRF and
  * area of fibrosis less than 50% of the lesion area.
* CNV membrane confirmed by presence of active leakage from the area of CNV seen by fluorescein angiography (FA) and color fundus photography (CFP) and at least two of the following items:

  * Drusen
  * Retinal Pigment Epithelium (RPE)-Atrophy
  * Exudates
  * Subretinal or intraretinal haemorrhage
* BCVA scores at both screening and baseline must be 23 letters or more as measured by the ETDRS-like charts (or approximate Snellen equivalent to 20/320).

Exclusion Criteria:

General:

* Inability to comply with study or follow-up procedures.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, not using or not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the Investigator in individual cases. (Female participants who are surgically sterilised/hysterectomised, or post-menopausal for longer than 2 years are not considered as being of child-bearing potential.)
* Any type of systemic disease or its treatment, in the opinion of the Investigator, including any medical condition (controlled or uncontrolled) that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk.
* Stroke or myocardial infarction less than 3 months prior to the date of informed consent signature.
* Uncontrolled blood pressure defined as systolic value of >160 mmHg or diastolic value of >100 mmHg at screening or baseline.
* Known hypersensitivity to aflibercept or any component of the aflibercept formulation, or fluorescein.
* Prior or current use of any systemic anti-VEGF drugs [e.g., bevacizumab (Avastin®) or ranibizumab (Lucentis®)].
* Current or planned use of systemic medications known to be toxic to the lens, retina or optic nerve, including chloroquine/hydroxychloroquine (Plaquenil®), deferoxamine, phenothiazines, tamoxifen, and ethambutol.
* Use of systemic or intravitreal corticosteroids for at least 30 consecutive days within 3 months prior to the date of informed consent signature.
* Use of other investigational drugs within 6 months prior to the date of informed consent signature.
* Patient was previously screened for participation in the study and was a screen failure.

Study eye:

* Any active periocular or ocular infection or inflammation (e.g., blepharitis, conjunctivitis, keratitis,scleritis, uveitis, endophthalmitis) at the time of screening or baseline.
* Uncontrolled glaucoma [intraocular pressure (IOP) ≥30 mmHg on medication or according to Investigator's judgment] at the time of screening or baseline.
* Neovascularisation of the iris or neovascular glaucoma at the time of screening or baseline.
* Inability of obtaining SD-OCT images of sufficient quality to be analysed.
* Any intraocular procedure (including Yttrium-Aluminum-Garnet capsulotomy) within 2 months prior to the date of informed consent signature or anticipated within the next 6 months following the date of informed consent signature.
* Visually significant cataract, aphakia, pseudoexfoliation glaucoma, vitreous haemorrhage, rhegmatogenous retinal detachment, proliferative diabetic retinopathy or CNV of any cause other than wAMD at the time of screening and baseline.
* Structural damage within 0.5 disc diameter of the centre of the macula at the time of screening or baseline that in the Investigator's opinion could preclude visual function improvement with treatment.
* Subretinal hemorrhage involving the central foveal subfield with a site of ≥1 disc diameter at the time of screening or baseline.
* Intraocular treatment with any anti-VEGF drug or intravitreal corticosteroids or previous treatment with photodynamic therapy or retinal laser therapy prior to the date of informed consent signature.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 patients will be recruited to this study, with approximately 75 randomised to each study arm (relaxed and strict retinal fluid treatment regimen). Assuming an approximate 20% screen failure rate, approximately 188 patients will need to be screened to have 150 patients found eligible and commencing treatment in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-12; Primary Completion 2022-03 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Change in best corrected visual acuity (BCVA) from baseline to end of treatment (EOS) at week 104. The primary outcome of the trial is the difference between the two arms in the mean change in BCVA from baseline to EOS. | From baseline to 24 months
  Change of BCVA from baseline to end of study at week 104

SECONDARY OUTCOMES:
The difference between the two arms in the mean change in BCVA from baseline to week 52. | From baseline to 24 months
The difference between the two arms in the mean change in central retinal thickness (CRT) from baseline to week 52 and to EOS. | From baseline to 24 months
The difference between the two arms in the mean number of injections from baseline to week 52 and to EOS. | From baseline to 24 months
The difference between the two arms in the proportion of patients showing newly developed geographic atrophy at week 52 and at EOS as compared to baseline. | From baseline to 24 months
The difference between the two arms in the mean change in the area of new and existing geographic atrophy from baseline to week 52 and to EOS. | From baseline to 24 months
The difference between the two arms in the proportion of patients showing no IRF and no SRF at week 52 and at EOS. | From baseline to 24 months
The difference between the two arms in the proportion of patients showing no SRF at week 52 and at EOS. | From baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, MD, PhD, Study Chair — Inselspital Bern, Department of Ophthalmology
Locations (2):
- Switzerland (2):
  - Department of Ophthalmology, University Hospital Bern, Bern
  - Inselspital Bern, Department of Ophthalmology, Bern